CLINICAL TRIAL: NCT00218179
Title: Prostate, Lung, Colon, and Ovarian Cancer (PLCO) Screen Trial
Brief Title: Assessing the Link Between Smoke Carcinogen Biomarkers and Lung Cancer Risk - 1
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: NIDA-13333-1; P50DA013333 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Tobacco Use Disorder; Lung Cancer
Keywords: Lung Cancer; Cotinine; NNAL; Carcinogens; Case-control; SNPs
MeSH Terms: conditions — Tobacco Use Disorder; Lung Neoplasms | interventions — 4-((methylnitrosoamino)-1-(3-pyridyl)but-1-yl)beta-omega-glucosiduronic acid; phenanthrene tetraol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Lung cancer cases diagnosed prior to 2007 among baseline smokers in the PLCO
  Interventions: Other: Non-intervention
- Controls: Subjects without lung cancer among smokers at baseline in the PLCO study
  Interventions: Other: Non-intervention

INTERVENTIONS:
Other: Non-intervention — Measured total NNAL and PheT as biomarkers of exposure
  Other Names: NNAL-glucuronide, phenanthrene tetraol

SUMMARY:
Lung cancer is the leading cause of cancer death in the United States. Currently it remains impossible to predict which smokers will get cancer. Each puff of a cigarette delivers a mixture of over 60 known carcinogens. Biomarkers that quantify carcinogen levels and metabolism are a useful tool and available to use. The purpose of this study is to assess the link between tobacco smoke carcinogen biomarkers and the risk of developing lung cancer.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in the United States. Approximately 90% of lung cancer is caused by cigarette smoking. While most lung cancer cases occur in smokers or ex-smokers, only 15-25% of smokers will get lung cancer. Currently it remains impossible to predict which smokers will get cancer.

Each puff of a cigarette delivers, along with nicotine, a mixture of over 60 known carcinogens. Most of these carcinogens require metabolic activation before they can negatively affect cell DNA and cause cancer. Biomarkers that quantify carcinogen levels and metabolic activity of carcinogens are a useful tool and available to use. The purpose of this study is to assess the link between tobacco smoke carcinogen biomarkers and the risk of developing lung cancer.

This observational case-control study will involve a random selection from a group of smokers who are participating in the Prostrate, Lung, Colon, and Ovarian Cancer (PLCO) Screen Trial. The chosen cases will include 300 incident lung cancer cases and 300 controls (participants who have had no diagnosis of lung cancer). Demographic and baseline data from the PLCO database will be obtained. Prior baseline blood samples from the PLCO trial will be obtained as well. Based on age, sex, and smoking history, participants will be grouped into triplets in order to pool their blood samples. These samples will then be analyzed to determine whether distributions of biomarker levels in lung cancer participants differ from those in non-lung cancer participants. This study will not involve recruitment of any participants, as data and samples from the PLCO trial will be used and no new blood samples will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Screening arm participants in the Prostate, Lung, Colon, and Ovarian Screen Trial (PLCO)
* Reported smoking on baseline questionnaire of PLCO
* Contributed biorepository samples

Exclusion Criteria:

* Unstable physical or mental health

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case-control study nested within the Prostate Lung Colorectal and Ovarian Cancer Screening Trial. Subjects consisted of screening arm subjects who were smokers at baseline and who contributed biorepository samples at the first screening visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Lung cancer | Cumulative incidence

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Church, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Church TR, Haznadar M, Geisser MS, Anderson KE, Caporaso NE, Le C, Abdullah SB, Hecht SS, Oken MM, Van Ness B. Interaction of CYP1B1, cigarette-smoke carcinogen metabolism, and lung cancer risk. Int J Mol Epidemiol Genet. 2010 Aug 5;1(4):295-309. PMID 21532841
- [Result] Church TR, Anderson KE, Caporaso NE, Geisser MS, Le CT, Zhang Y, Benoit AR, Carmella SG, Hecht SS. A prospectively measured serum biomarker for a tobacco-specific carcinogen and lung cancer in smokers. Cancer Epidemiol Biomarkers Prev. 2009 Jan;18(1):260-6. doi: 10.1158/1055-9965.EPI-08-0718. PMID 19124507
- [Result] Fang G, Haznadar M, Wang W, Yu H, Steinbach M, Church TR, Oetting WS, Van Ness B, Kumar V. High-order SNP combinations associated with complex diseases: efficient discovery, statistical power and functional interactions. PLoS One. 2012;7(4):e33531. doi: 10.1371/journal.pone.0033531. Epub 2012 Apr 19. PMID 22536319